CLINICAL TRIAL: NCT04834739
Title: Comparison of Functional Capacities of Healthcare Workers With and Without Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 208
Record Dates: First submitted 2021-01-10; First posted 2021-04-08 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Functional Capacity
Keywords: Covid-19; healthcare worker; functional capacity
MeSH Terms: conditions — COVID-19 | interventions — antigens, CD200

STUDY DESIGN:
Intervention Model Description: 30 volunteer healthcare workers who had Covid-19 and stayed in hospital or at home were included. In control group, 30 volunteer healthcare workers who were matched for age and gender with study group were included and these persons had not have Covid-19. Healthcare workers who have had Covid-19 disease will be evaluated for the first time within 1 month after their diagnosis with RT-PCR test for SARS-CoV-2 (The condition of completing isolation process of the patients will be sought).
Who Masked: Outcomes Assessor
Masking Description: study and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (30 volunteer healthcare workers who had Covid-19 (Active Comparator): 30 volunteer healthcare workers who had Covid-19 and stayed in hospital or at home were included.
  Interventions: Other: 6 minute walk test; Other: 1 minute Sit to Stand Test; Other: Fatigue Severity Scale; Other: Medical Research Council (MRC) dyspnea scale; Other: SF-12; Other: Beck Depression Inventory; Other: Beck Anxiety Inventory; Other: 5 times sit to stand test; Other: 6 point Likert Scale
- Control group (30 volunteer healthcare workers who had not have Covid-19) (Active Comparator): In control group, 30 volunteer healthcare workers who were matched for age ande gender with study group were included and these persons had not have Covid-19.
  Interventions: Other: 6 minute walk test; Other: 1 minute Sit to Stand Test; Other: Fatigue Severity Scale; Other: Medical Research Council (MRC) dyspnea scale; Other: SF-12; Other: Beck Depression Inventory; Other: Beck Anxiety Inventory; Other: 5 times sit to stand test; Other: 6 point Likert Scale

INTERVENTIONS:
Other: 6 minute walk test — The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. 30 m long corridor is used for this test .
Other: 1 minute Sit to Stand Test — The 1-minute STS test is performed with a chair of standard height of 46 cm without arm rests. The patient should be ensured to be seated upright on the chair positioned against a wall. The patient sat with the knees and hips flexed to 90°, feet placed flat on the floor hip-width apart, and the hands placed on the hips.The number of repetitions is measured.
Other: Fatigue Severity Scale — The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders
Other: Medical Research Council (MRC) dyspnea scale — The MRC dyspnea scale is a questionnaire that consists of five statements about perceived breathlessness: grade 1, "I only get breathless with strenuous exercise"; grade 2, "I get short of breath when hurrying on the level or up a slight hill"; grade 3, "I walk slower than people of the same age on the level because of breathlessness or have to stop for breath when walking at my own pace on the level"; grade 4, "I stop for breath after walking 100 yards or after a few minutes on the level"; grade 5, " I am too breathless to leave the house".
Other: SF-12 — The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
Other: Beck Depression Inventory — The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression
Other: Beck Anxiety Inventory — Beck Anxiety Scale is a 21-item, internationally valid, self-report rating inventory that measures the anxiety level.
Other: 5 times sit to stand test — The 5XSST scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times. The equipment need in performing 5XSST test includes: Stopwatch and standard height chair with straight back (43-45 cm, 17-18 inches high). Then the instruction is given by asking the test taker to sit on the chair by resting their back. Also, the test taker is instructed to fold their arms across their chest. Then the test taker should be instructed to do sit-to-stand five times, as quickly as possible, at the count of go and without their back or leg resting on the chair between the interval of repetition.
Other: 6 point Likert Scale — Job performance was assessed by asking "How do you evaluate your job performance?" on 6-point Likert scale.A 6 point likert scale forces choice and gives better data.The 6 point Likert scale offers options for ''Excellent, very good, good, fair, poor and very poor''. 6 point scale anges from 1(very poor) to 5 (excellent).

SUMMARY:
This study aimed to investigate if the functional capacity of health workers sustained covid 19 infection effects functional capacity , quality of life and mood of health workers when comparing healthy health workers.

DETAILED DESCRIPTION:
This study was designed in Physical Medicine and Rehabilitation Service of Gaziosmanpasa Training and Research Hospital between January 4 and June 30, 2021.Data of the health workers from our hospital who suffered from Covid-19 disease and matched control group who had not have Covid-19 disease participants were analyzed. Participants signed a general consent .Inclusion criteria; being a health worker over the age of 18 (for both groups), having had SARS-CoV-2 (Covid 19) disease for last 1 month and completed the isolation process, volunteer to participate in the study, , being able to walk or sit and stand without any help, speaking and understand Turkish language. Exclusion criteria (for both study and control group); Neurological or musculoskeletal disease that causes gait impairment, cognitive impairment, having unstable cardiac, respiratory and metabolic disease.(The first assessment will be made within the 1st month after the patient's Covid 19 positivity is detected; control will be made three times in the 2nd, 4th and 6 months)

30 volunteer healthcare workers who had Covid-19 were included to study group. 30 age and gender matched volunteer healthcare workers were included to control group. Healthcare workers who have had Covid-19 disease will be evaluated for the first time within 1 month after their diagnosis with RT-PCR test for SARS-CoV-2.

Symptom questioning will be reported including the initial symptoms of Covid-19 and ongoing complaints of the patients. During the examination, muscle strength will be evaluated by the Medical Research Council (MRC) total score. Resting heart rate, blood pressure and oxygen saturation (by pulse oxymeter) measurement will be applied to both groups before and after the following tests: 1-min sit-to-stand (1MSTS) test, 5 times sit-to-stand (5TSTS) test, 6 minutes walk test (6MWT).

MRC dyspnea scale will be performed as a measure of patient's complaint of shortness of breath,Job performance was assessed by asking "How do you evaluate your job performance?" on 6-point Likert scale, Short Form-12 (Short Form 12, SF-12) will be used to assess quality of life, mood disorder wil be measured by Beck Anxiety Inventory and Beck Depression Inventory, Fatigue severity scale(FSS) will be performed as level of fatigue. The first evaluation wil be made within 1 month after one positive RT-PCR test for SARS-CoV-2 is detected; control evaluations will be made in the 2nd, 4th and 6th months after positivity of RT-PCR test for SARS-CoV-2. Finally, the patient's sex, age, body mass index (BMI), height, education status, career, status of hospitalization, length of hospitalization, comorbidities , pulmonary involvement that diagnosed radiological methods and examination of symptoms related with Covid-19 will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being a health worker over the age of 18 (for both control group)
* Having had SARS-CoV-2 (Covid 19) disease in the last 1 month and completed the isolation process
* Volunteer to participate in the study, being discharged from the hospital and completing the isolation process at home (The first assessment will be made within the 1st month after the patient's Covid 19 positivity is detected; control will be made three times in the 2nd, 4th and 6th months)
* Being able to walk or sit and stand without any help
* Speaking and understand the Turkish language.

Exclusion Criteria:*For both study and control group

* Neurological or musculoskeletal disease that causes gait impairment
* Cognitive impairment
* Having unstable cardiac, respiratory and metabolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
1 minute sit to stand test | Change at 2nd, 4th and 6th months.
  1 minute sit to stand test will be used to measure aerobic capacity and endurance.
5 times sit to stand test | Change at 2nd, 4th and 6th months.
  The five Times Sit to Stand Test (5x Sit-To-Stand Test) commonly abbreviated as 5XSST is used to assesses functional lower extremity strength, transitional movements, balance, and fall risk in older adults
6 minute walk test | Change at 2nd, 4th and 6th months.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

SECONDARY OUTCOMES:
Medical Research Council (MRC) dyspnea scale | Change at 2nd, 4th and 6th months
  Medical Research Council (MRC) dyspnea scale is a questionnaire that consists of five statements about perceived breathlessness in dailt activities.
6 point Likert Scale | Change at 2nd, 4th and 6th months.
  Job performance was assessed by asking "How do you evaluate your job performance?" on 6-point Likert scale.
Fatigue Severity Scale | Change at 2nd, 4th and 6th months.
  The Fatigue Severity Scale is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders.
Beck Depression Inventory | Change at 2nd, 4th and 6th months.
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression
Beck Anxiety Scale | Change at 2nd, 4th and 6th months.
  Beck Anxiety Scale is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults
Short form 12 | Change at 2nd, 4th and 6th months.
  Short form 12 will be used to measure quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yilmaz Yalcinkaya, 3, Study Chair — University of Health Science,Gaziosmanpasa Training and Research Hospital; Ozden Ozyemisci Taskiran, 4, Study Director — Koç University
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)